CLINICAL TRIAL: NCT03746548
Title: Audiological Benefit and Quality of Life With Two Bone Conduction Systems: ADHEAR vs. Contact Mini
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dominik Riss (Other)
Responsible Party: Sponsor-Investigator, Dominik Riss, Assoc. Prof. PD. Dr., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1573/2017
Record Dates: First submitted 2018-11-11; First posted 2018-11-19 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Conductive Hearing Loss
MeSH Terms: conditions — Hearing Loss, Conductive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CM-ADHEAR (Other): First patients use the Contact Mini (conventional bone conduction device used with a soft band or headband) then ADHEAR (adhesive bone conduction device)
  Interventions: Device: Adhear; Device: Contact Mini (CM)
- ADHEAR - CM (Other): First patients use ADHEAR (adhesive bone conduction device) then CM (conventional bone conduction device used with a soft band or headband)
  Interventions: Device: Adhear; Device: Contact Mini (CM)

INTERVENTIONS:
Device: Adhear — Patients are wearing the Adhesive bone conduction hearing device (Adhear) for 2 weeks
Device: Contact Mini (CM) — Patients are wearing the Conventional bone conduction hearing device (Contact Mini) for 2 weeks

SUMMARY:
Patients with conductive hearing loss fitting the inclusion criteria will be asked to participate in the study. All subjects will be randomized to wear either first the adhesive or the conventional bone conduction hearing aid. They will wear either device for two weeks. They will use the second device for another two weeks. Audiologic tests and quality of life questionnaires will be assessed at the beginning of the study after two weeks with the first device and after two weeks with the second device. Additionally, all patients will be asked to keep a diary including daily wearing time of the device.

DETAILED DESCRIPTION:
The primary objective of this study is to show, that the ADHEAR will be worn ~75%(~11 to 15 hours per day) of the waking hours, whereas the Contact Mini will be worn ~ 50% (~5 - 8 hours per day) of the waking hours (p<0.05). The authors expect this difference due to increased wearing comfort, reduced/no pressure to the skin of the ADHEAR. The primary objective will be assessed with the diary patients are asked to use.

Audiologic testing will consist of free field audiometry, Freiburger monosyllables test and Oldenburg sentence test. All tests will be performed with and without the devices.

Quality of life and hearing related questionnaires will consist of the AQoL-8D and the SSQ12.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria

  * Unilateral and/or bilateral conductive hearing loss (CHL)
  * The bone conduction threshold for the patient's affected ear shall be better than or equal to 25 dB HL (PTA BC for 0.5, 1, 2, 3 kHz).
  * Subjects aged 13 years or older
  * Capable of the German language
  * Willingness and ability to perform all tests required for the study
  * Signed, and dated informed consent before the start of any study specific procedure

Exclusion Criteria:

Exclusion criteria

* Pregnancy or breastfeeding
* Patient is intolerant of the materials as described by Manufacturer's IFU
* Patient presents with a skin or scalp condition that may preclude the attachment of the adhesive adapter.
* Patient cannot perform the audiological tests or is unable to fill out the questionnaires.
* Patient presents with retrocochlear, or central auditory disorder.
* any physical, psychological, or emotional disorder that would interfere with the ability to perform on test and rehabilitation procedures

Ages: 13 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Wearing time | 1 year
  Wearing time per day of the two devices

CONTACTS AND LOCATIONS:
Locations (1):
- MUW AKH, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No